CLINICAL TRIAL: NCT01721629
Title: Weaning of Nasal Continuous Positive Airway Pressure in Infants Born With a Gestational Age Under 32 Weeks: a Randomized Controlled Multicenter Trial
Brief Title: Weaning of Nasal Continuous Positive Airway Pressure (CPAP) in Premature Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aarhus University Hospital (Other)
Responsible Party: Principal Investigator, Christina Friis Jensen, MD, Ph.D. student, Aarhus University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AAUH190280
Record Dates: First submitted 2012-09-25; First posted 2012-11-06 (Estimated); Last update posted 2017-05-01 (Actual); Status verified 2017-04

CONDITIONS: Prematurity; Respiratory Distress Syndrome, Infant
Keywords: Nasal cpap weaning; Premature infants; Respiratory distress syndrome; Randomized controlled trial
MeSH Terms: conditions — Premature Birth; Respiratory Distress Syndrome, Newborn; Respiratory Distress Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sudden wean of nasal CPAP (Other): The CPAP is taken off at the morning ward round. If the discontinuation of the CPAP fails according to prespecified failure criteria, CPAP is recommenced and continued for at least 24 hours. Then a new evaluation takes place and if the infant again meets the inclusion criteria another attempt of sudden wean can be undertaken. Infants are considered successfully weaned if they are off CPAP for three days.
  Interventions: Procedure: Sudden wean of nasal CPAP
- Gradual wean of nasal CPAP pressure (Other): The reduction of the CPAP pressure begins at the morning ward round and the pressure is reduced in steps with 1 cmH2O maximum once a day. Each time the pressure is to be reduced the infant needs to be evaluated according to the inclusion criteria and only if these are still met, will the pressure be reduced. When a CPAP pressure at 4 cmH2O is reached the infant is treated with this pressure for 24 hours and then the CPAP is discontinued. Infants are considered successfully weaned if they are off CPAP for three days.
  Interventions: Procedure: Gradual wean of nasal CPAP

INTERVENTIONS:
Procedure: Sudden wean of nasal CPAP
  Arms: Sudden wean of nasal CPAP
Procedure: Gradual wean of nasal CPAP
  Arms: Gradual wean of nasal CPAP pressure

SUMMARY:
The aim of this study is to investigate two different strategies for the withdrawal of CPAP in preterm infants born before 32 weeks of gestation.

ELIGIBILITY:
Inclusion Criteria:

* Gestational age < 32 weeks at birth
* Current gestational age > 28+6 weeks
* Nasal CPAP for > 24 hours
* Nasal CPAP pressure < 8 cmH2O
* Oxygen requirement < 30% and not increasing
* Respiratory rate < 70 per minute
* Less than 3 episodes of oxygen saturation < 70% or a heart rate < 70 beat per minute in the preceding 24 hours
* Tolerates time off CPAP during cares (up to 15 minutes)

Exclusion Criteria:

* Congenital malformations of the heart (except patent ductus arteriosus, atrial septal defect and patent foramen ovale), lung, and gastrointestinal tract
* Surgical procedures performed on the gastrointestinal tract
* Known or suspected to have congenital neuromuscular disease
* Known or suspected syndrome

Max Age: 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 380 (Actual)
Dates: Start 2012-09; Primary Completion 2017-04-28 (Actual); Study Completion 2017-04-28 (Actual)

PRIMARY OUTCOMES:
Weight at a gestational age of 40 weeks | Up to 16 weeks

SECONDARY OUTCOMES:
Weight at completed withdrawal of nasal CPAP | From date of birth until the date of complete withdrawal of nasal CPAP. Expected median of 14 days
Duration of oxygen treatment | Up to 6 months
Duration of nasal CPAP therapy | Up to 6 months
Length of stay in the hospital | Expected median 54 days
Occurence of bronchopulmonary dysplasia | Up to 12 weeks
  The occurrence of bronchopulmonary dysplasia is defined as need for oxygen therapy (> 21%) at a gestational age of 36 weeks or treatment with oxygen > 21% for at least 28 days (a day of treatment with oxygen > 21% means that the infant received oxygen > 21% for more than 12 hours that days)
Parental anxiety | Up to 6 months
Depression in parents | Up to 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Christina F Jensen, MD, Principal Investigator — The Perinatal Epidemiology Research Unit and Department of Paediatrics, Aarhus University Hospital; Tine B Henriksen, Professor, Study Director — Department of Paediatrics, Aarhus University Hospital; Kirsten Wisborg, Centre Director, DMSc, Study Chair — Aarhus University Hospital, Head-Neuro Centre; Finn Ebbesen, Professor, Study Chair — Department of Paediatrics, Aalborg University Hospital; Anna S Sørensen, MD, Ph.D., Study Chair — The Perinatal Epidemiology Research Unit and Department of Paediatrics, Aarhus University Hospital
Locations (6):
- Denmark (6):
  - Aalborg University Hospital, Department of Pediatrics, Aalborg, DK
  - Aarhus University Hospital, Department of Pediatrics, Aarhus, DK
  - Herning Hospital, Department of Pediatrics, Herning, DK
  - Viborg Hospital, Department of Pediatrics, Viborg, DK
  - Vendsyssel Hospital, Department of Pediatrics, Hjørring
  - Randers Hospital, Department of Pediatrics, Randers

REFERENCES:
- [Derived] Jensen CF, Sellmer A, Ebbesen F, Cipliene R, Johansen A, Hansen RM, Nielsen JP, Nikitina OH, Petersen JP, Henriksen TB. Sudden vs Pressure Wean From Nasal Continuous Positive Airway Pressure in Infants Born Before 32 Weeks of Gestation: A Randomized Clinical Trial. JAMA Pediatr. 2018 Sep 1;172(9):824-831. doi: 10.1001/jamapediatrics.2018.2074. PMID 30039171